CLINICAL TRIAL: NCT01444898
Title: Effects of Exenatide on Obesity and Appetite in Overweight Patients With Prader-Willi Syndrome
Brief Title: Effects of Exenatide on Overweight Adolescents With Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Mitchell E. Geffner, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI 11-00227
Record Dates: First submitted 2011-09-27; First posted 2011-10-03 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Obesity; Weight; Exenatide; Byetta; Pediatrics; Adolescents
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity; Body Weight | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exenatide (Experimental): All subjects enrolled in this study will be given Exenatide for 6 months. Exenatide: The investigators will give patients naive to GLP-1 agonists exenatide per manufacturer dosing recommendations for 6 months. The investigators will begin by giving 5 mcg subcutaneously twice a day for 1 month and then increase the dose to 10 mcg subcutaneously twice a day for the remainder of the study (5 months).
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — The investigators will give patients naive to GLP-1 agonists exenatide per manufacturer dosing recommendations for 6 months. The investigators will begin by giving 5 mcg subcutaneously twice a day for 1 month and then increase the dose to 10 mcg subcutaneously twice a day for the remainder of the study (5 months).
  Other Names: Byetta

SUMMARY:
Prader-Willi Syndrome (PWS) is one of the most common genetic causes of obesity. Obesity is a major source of morbidity and mortality in this population. It can lead to sleep apnea, cor pulmonale, diabetes mellitus, and atherosclerosis. PWS has distinct characteristics that set it apart from other forms of obesity including insatiable appetite and food-seeking behavior which can be disruptive to home and school activities, and can cause severe social and psychological turmoil within families. PWS is also associated with unique hormonal abnormalities, most notably hyperghrelinemia. Ghrelin is a gut hormone produced in the stomach that stimulates food intake during a fast. It is hypothesized that the extremely high ghrelin levels in patients with PWS may cause or contribute to their insatiable appetite. Exenatide, a medication used in the treatment of type 2 diabetes mellitus in adults, appears to suppress ghrelin levels and cause weight loss. It was designed to mimic glucagon-like peptide 1 (GLP-1), an incretin hormone that stimulates insulin secretion and delays gastric emptying, among other effects. In the present study, the investigators will investigate the effects of a 6 month trial of exenatide in overweight adolescents with PWS. The investigators will quantify the changes in weight and body composition, as well as subjective measures of appetite, and concentrations of appetite-associated hormones. The investigators hypothesize that exenatide will improve weight, body composition, appetite, and plasma ghrelin levels during the treatment period.

DETAILED DESCRIPTION:
BACKGROUND:

Prader-Willi syndrome (PWS) is associated with hyperphagia and hyperghrelinemia with major morbidity because of obesity without effective medical treatment targeting hyperphagia. Exenatide (Byetta [synthetic Exendin-4]; AstraZeneca, Wilmington DE) is a GLP-1 receptor agonist which reduces appetite and weight and may be an effective treatment in PWS.

OBJECTIVE: The objective of this study is to determine the effect of a 6-month trial of exenatide on appetite, weight and gut hormones in youth with PWS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Prader Willi Syndrome confirmed by genetic testing (DNA methylation or FISH)
* Ages 13-20 years
* body mass index (BMI) > 85th percentile for age and gender

Exclusion Criteria:

* Is currently using or has previously used a glucagon-like peptide-1 (GLP-1) agonist
* History of pancreatitis, or renal failure
* History of familial pancreatitis
* Amylase, or lipase levels > 2.5 times the upper limit of normal any time in the previous 2 years
* Creatinine clearance < 30 mL/min
* Other syndromic diagnoses
* gastrointestinal (GI) or renal illness in the 1 month prior to entering study
* Inability to take study drug
* Pregnancy
* Initiation of growth hormone (GH), estrogen, or testosterone or change > 25% of dose/kg/day during the 6 months prior to starting study
* Non-English speaking

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Jeandron, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstone AP. The hypothalamus, hormones, and hunger: alterations in human obesity and illness. Prog Brain Res. 2006;153:57-73. doi: 10.1016/S0079-6123(06)53003-1. PMID 16876568
- [Background] Goldstone AP. Prader-Willi syndrome: advances in genetics, pathophysiology and treatment. Trends Endocrinol Metab. 2004 Jan-Feb;15(1):12-20. doi: 10.1016/j.tem.2003.11.003. PMID 14693421
- [Background] Suzuki K, Simpson KA, Minnion JS, Shillito JC, Bloom SR. The role of gut hormones and the hypothalamus in appetite regulation. Endocr J. 2010;57(5):359-72. doi: 10.1507/endocrj.k10e-077. Epub 2010 Apr 14. PMID 20424341
- [Background] Wren AM, Seal LJ, Cohen MA, Brynes AE, Frost GS, Murphy KG, Dhillo WS, Ghatei MA, Bloom SR. Ghrelin enhances appetite and increases food intake in humans. J Clin Endocrinol Metab. 2001 Dec;86(12):5992. doi: 10.1210/jcem.86.12.8111. PMID 11739476
- [Background] Cummings DE, Clement K, Purnell JQ, Vaisse C, Foster KE, Frayo RS, Schwartz MW, Basdevant A, Weigle DS. Elevated plasma ghrelin levels in Prader Willi syndrome. Nat Med. 2002 Jul;8(7):643-4. doi: 10.1038/nm0702-643. No abstract available. PMID 12091883
- [Background] Paik KH, Jin DK, Song SY, Lee JE, Ko SH, Song SM, Kim JS, Oh YJ, Kim SW, Lee SH, Kim SH, Kwon EK, Choe YH. Correlation between fasting plasma ghrelin levels and age, body mass index (BMI), BMI percentiles, and 24-hour plasma ghrelin profiles in Prader-Willi syndrome. J Clin Endocrinol Metab. 2004 Aug;89(8):3885-9. doi: 10.1210/jc.2003-032137. PMID 15292322
- [Background] Rosenstock J, Klaff LJ, Schwartz S, Northrup J, Holcombe JH, Wilhelm K, Trautmann M. Effects of exenatide and lifestyle modification on body weight and glucose tolerance in obese subjects with and without pre-diabetes. Diabetes Care. 2010 Jun;33(6):1173-5. doi: 10.2337/dc09-1203. Epub 2010 Mar 23. PMID 20332357
- [Background] Perez-Tilve D, Gonzalez-Matias L, Alvarez-Crespo M, Leiras R, Tovar S, Dieguez C, Mallo F. Exendin-4 potently decreases ghrelin levels in fasting rats. Diabetes. 2007 Jan;56(1):143-51. doi: 10.2337/db05-0996. PMID 17192476
- [Background] Seetho IW, Jones G, Thomson GA, Fernando DJ. Treating diabetes mellitus in Prader-Willi syndrome with Exenatide. Diabetes Res Clin Pract. 2011 Apr;92(1):e1-2. doi: 10.1016/j.diabres.2010.12.009. Epub 2011 Jan 11. PMID 21227526
- [Result] Salehi P, Hsu I, Azen CG, Mittelman SD, Geffner ME, Jeandron D. Effects of exenatide on weight and appetite in overweight adolescents and young adults with Prader-Willi syndrome. Pediatr Obes. 2017 Jun;12(3):221-228. doi: 10.1111/ijpo.12131. Epub 2016 Apr 13. PMID 27071367

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide: All subjects enrolled in this study will be given Exenatide for 6 months. The investigators will give patients naive to GLP-1 agonists exenatide per manufacturer dosing recommendations for 6 months. The investigators will begin by giving 5 mcg subcutaneously twice a day for 1 month and then increase the dose to 10 mcg subcutaneously twice a day for the remainder of the study (5 months).
Period: Overall Study
Arm/Group | Exenatide
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [14.7 to 24.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Region of Enrollment = California
  participants
    United States | 10
Weight [Mean (Standard Deviation); unit: kg] — Weight (kg)
  kg | 102.5 (18.6)
BMI [Median (Inter-Quartile Range); unit: kg m^-2] — BMI (kg m^-2)
  kg m^-2 | 41.7 [34.1 to 55]
BMI Z-Score [Mean (Standard Deviation); unit: units on a scale] | 3.5 (1.1)
Glycosylated hemoglobin (HbA1c) [Median (Inter-Quartile Range); unit: percentage of total hemoglobin] — Glycosylated hemoglobin (HbA1c), percentage of total hemoglobin
  percentage of total hemoglobin | 5.9 [5.6 to 7.9]
Insulin [Median (Inter-Quartile Range); unit: uIU ml^-1] — Insulin (u/U ml^-1)
  uIU ml^-1 | 10.5 [6 to 21]
Leptin [Mean (Standard Deviation); unit: ng ml ^-1] — Leptin (ng ml ^-1)
  ng ml ^-1 | 36.4 (18.3)
Acy Ghr [Median (Inter-Quartile Range); unit: pg ml ^-1] — Acylated ghrelin, Acy Ghr (pg ml ^-1)
  pg ml ^-1 | 362.3 [259 to 740.7]
PP [Median (Inter-Quartile Range); unit: pg ml ^-1] — Pancreatic polypeptide, PP (pg ml ^-1)
  pg ml ^-1 | 89 [31 to 662]
Appetite [Mean (Standard Deviation); unit: units on a scale] — Appetite scores - For 1 and 2: 11 item questionnaire divided into subcategories of behavior (5 questions), drive (4 questions), severity (2 questions). Tallied and analyzed as total and subcategory scores. Each question scored 1-5 with higher scores correlating with worse hyperphagia.
  Possible ranges: Total 11-55, behavior 5-25, drive 4-20, severity 2-10
  units on a scale
    Total Appetite Score | 32.2 (8.7)
    Appetite Behavior | 14.5 (4.9)
    Appetite Drive | 12.6 (3.1)
    Appetite Severity | 5.1 (1.5)
Adiposity [Number; unit: percentage of fat] — Truncal fat as measured by dual x-ray absorptiometry
  percentage of fat | 44.7
Adiposity [Mean (Standard Deviation); unit: kg] — Mean truncal fat
  kg | 20 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight (kg) after 6 months of treatment with study drug. Described as mean +/- SD
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exenatide
Number analyzed (Participants) | 10
kg | -.5 (.9)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .07, Mixed Models Analysis

2. Primary Outcome: % Change in Body Mass Index (BMI)
Description: Prior to analysis, distributions were evaluated for normality and natural log transformation was performed to analyse data not normally distributed. Data are presented as mean ±SD unless not normally distributed, in which case they are presented as median with intra-quartile ranges (25th and 75th percentiles). Within-subject changes between visits were analysed by mixed model repeated measures. When the overall F-test for difference among visits was significant, Dunnett-adjusted pairwise comparisons were made between baseline and each subsequent visit.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in BMI
Arm/Group | Exenatide
Number analyzed (Participants) | 10
% change in BMI | 1.3 (2)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis

3. Primary Outcome: Change in BMI Z-Score
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exenatide
Number analyzed (Participants) | 10
units on a scale | .1 (.4)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .8, Mixed Models Analysis

4. Primary Outcome: Change in HbA1c (%)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Exenatide
Number analyzed (Participants) | 10
percentage | -.3 (.2)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .04, Mixed Models Analysis

5. Primary Outcome: Change in Insulin Levels
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: u/U ml^-1
Arm/Group | Exenatide
Number analyzed (Participants) | 10
u/U ml^-1 | 3 (.5)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .8, Mixed Models Analysis

6. Primary Outcome: Change in Leptin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng ml^-1
Arm/Group | Exenatide
Number analyzed (Participants) | 10
ng ml^-1 | -7.4 (3.8)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .2, Mixed Models Analysis

7. Primary Outcome: Change in Acy Ghr
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg ml^-1
Arm/Group | Exenatide
Number analyzed (Participants) | 10
pg ml^-1 | 263 (99.5)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .2, Mixed Models Analysis

8. Primary Outcome: Change in Pancreatic Peptide (PP)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg ml^-1
Arm/Group | Exenatide
Number analyzed (Participants) | 10
pg ml^-1 | 15 (6)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .04, Mixed Models Analysis

9. Primary Outcome: Appetite Scores
Description: Appetite scores using a syndrome-validated hyperphagia questionnaire
  11 item questionnaire divided into subcategories of behavior (5 questions), drive (4 questions), severity (2 questions). Tallied and analyzed as total and subcategory scores. Each question scored 1-5 with higher scores correlating with worse hyperphagia.
  Possible ranges: Total 11-55, behavior 5-25, drive 4-20, severity 2-10
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exenatide
Number analyzed (Participants) | 10
units on a scale
  Total Appetite Score Baseline | 32.2 (8.7)
  Total Appetite Score 6 month | 25.4 (7.2)
  Behavior Score Baseline | 14.5 (4.9)
  Behavior Score 6 months | 10.6 (3.8)
  Drive Score Baseline | 12.6 (3.1)
  Drive Score 6 months | 10.4 (2.7)
  Severity Score Baseline | 5.1 (1.5)
  Severity Score 6 months | 4.4 (2.2)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .004, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Exenatide
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=10)
abdominal discomfort with diarrhea (Gastrointestinal disorders) | 2 (2) — One subject reported abdominal cramping and diarrhea for a short period because of acute infectious gastroenteritis. Another subject experienced mild abdominal discomfort and diarrhea after doubling the dose of exenatide for 1 d.

LIMITATIONS AND CAVEATS:
* small sample size
* referral bias due to small recruitment area
* confounding factors during the study, including variations in eating schedule, psychotropic medications, caretaker supervision and activity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No